CLINICAL TRIAL: NCT06223152
Title: Evaluation of the Effectiveness of a Guidance Program for Parents of Deaf Children
Acronym: Irsa-Triangle
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: My collaborator on this study (valérie deville) is away for an extended period.
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRSA-Triangle Wallonie
Record Dates: First submitted 2022-06-20; First posted 2024-01-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Deaf Nonspeaking, Not Elsewhere Classified
Keywords: deaf children; communication; language parental support
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- deaf children and parents (Experimental)
  Interventions: Other: parental support

INTERVENTIONS:
Other: parental support — parental support

SUMMARY:
The purpose of this project is to evaluate the effectiveness of a parent guidance program on (1) the parent's communication skills, (2) the parent's sense of competence and (3) the child's language development. Concretely, 11 guidance sessions will be offered to parents by alternating two group sessions (in a common place) and one family session (at home). These sessions will be given every week and will last approximately 2 hours. The sessions will focus on working on and learning adult attitudes conducive to the development of communication and language in the child. These sessions will be interactive through questions (wooclap), exchanges, video illustrations, role playing, etc. A practical application will be proposed in daily life with the help of the video-feedback technique during the home sessions, individually with the parent.

The effectiveness of this intervention will be evaluated via a pre- and post-test conducted in the families' homes. Episodes of parent-child interactions in a play situation will be filmed and coded in order to assess the parents' communication skills (receptivity, reactivity, language support strategies, etc.). The feeling of parental competence as well as the child's language will be estimated using parent questionnaires.

The investigators hypothesize that parent guidance sessions will have an effect on the communication skills of parents of deaf children and will indirectly improve their sense of parenting competence as well as the child's language development. This study will therefore offer avenues for adapting the support of families of deaf children.

ELIGIBILITY:
Inclusion Criteria:

* deaf children and parents
* 18 months - 4 years

Exclusion Criteria:

-

Ages: 18 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Communication between parent and child | troughout the entire study, an average of 40 months
  An episode of parent-child interactions in a play situation will be filmed before and after the intervention (pre- and post-test) in order to assess parents' communicative skills (receptivity, responsiveness, language support strategies, etc.). Fifteen minutes of free face-to-face play with a common material (Fischer Price's farm) will be recorded to provide a sample of parent-child interaction in a natural situation.
  The filmed interactions will be coded qualitatively via coding of verbal, paraverbal, and non-verbal exchanges that will be done using an analysis/observation grid created based on a grouping of elements from different existing grids (Adams, Gaile, Freed & Lockton, 2011; Ducerf, 2013; Prutting & Kirchner, 1987, Sylvestre, A. et al, 2019).
Child's language development | troughout the entire study, an average of 40 months
  Questionnaire estimating the child's language development French Inventory of Communication Development (Kern, Langue, Zesigner, & Bovet, 2010)
Questionnaires assessing the feeling of parental competence | troughout the entire study, an average of 40 months
  Global Scale of Sense of Parental Competence (GSSPC) (Meunier & Roskam, 2009) Adaptation of the SPISE-R, Scale of Parental Involvement and Self-Efficacy, revised (DesJardin, 2020)

CONTACTS AND LOCATIONS:
Locations (1):
- Bragard, Louvain-la-Neuve, Belgium